CLINICAL TRIAL: NCT07149116
Title: Intratracheal Sealing of Tracheostomy Immediately After Decannulation
Brief Title: Intratracheal Tracheostomy Sealing - A Clinical Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-112-22
Record Dates: First submitted 2025-08-08; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Tracheostomy Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intratracheal sealing disc (Experimental): A silicone disc is inserted through the tracheostomy to seal it. The disc is removed through the remaining tracheostomy once the wound has healed around it.
  Interventions: Device: Tracheostomy sealing

INTERVENTIONS:
Device: Tracheostomy sealing — A non-classified silicone-based prototype device designed to temporarily seal the tracheostomy tract from within the airway for up to 7 days after decannulation.

SUMMARY:
The purpose of this study is to investigate a new treatment method for tracheostomies - the term for the opening you have in your neck.

The treatment method seals the stoma tract from within the trachea. The aim is to improve lung function and voice quality, as well as to promote wound healing.

Study procedure: A silicone sealing device will be inserted into the stoma tract. This may cause temporary discomfort around the site and may induce some coughing. You will then undergo a pulmonary function test - also known as a spirometry test.

For the following 7 days, the sealing device will remain in the stoma tract and provide an airtight seal. You will be examined daily with spirometry, and the healing of the stoma tract will be closely monitored. A member of the research team will be present with you around the clock to ensure that the device remains correctly positioned. This is a safety precaution in the unlikely event that the sealing device dislocates into the airway.

After 7 days, the sealing device will be removed through the nearly healed stoma tract simply by pulling it out. This may again cause slight irritation or coughing.

DETAILED DESCRIPTION:
Background Tracheostomy is a surgical opening in the airway, most commonly performed as part of mechanical ventilation therapy.

It is the most frequently performed surgical procedure in critically ill patients admitted to intensive care units (ICUs) worldwide.

Based on the background literature, we estimate that approximately 1 million tracheostomies are performed globally each year.

An international study found that 24% of ventilated ICU patients were treated through a tracheostomy.

A tracheostomy is formed by creating an open channel from the trachea to the skin surface, typically located just above the sternum. The tract is kept open using a tracheostomy cannula, through which the patient breathes.

The indication for tracheostomy is most often a need for prolonged mechanical ventilation or upper airway obstruction at the level of the larynx due to tumour or scarring following surgery or radiotherapy.

Current Treatment When the patient no longer requires the tracheostomy, the cannula is removed (a process known as decannulation), and the tracheostomy site is covered with an adhesive dressing.

This dressing-based approach is associated with significant air leakage from the airway, which compromises speech, cough strength, airway clearance, and general pulmonary rehabilitation following ventilator therapy.

The Problem The cough mechanism is crucial for maintaining alveolar patency and thereby ensuring ventilation of all lung regions.

If alveoli collapse due to secretion retention or insufficient airway pressure, the risk of pneumonia and inadequate pulmonary function increases significantly-potentially to a degree necessitating reintubation.

During a cough, the glottis closes, and pressure builds within the lungs. Upon glottic opening, this pressure is released, aiding the reopening of collapsed lung segments.

Normal lung physiology and effective coughing depend on an airtight airway, where all airflow passes through the vocal cords and larynx once the glottis opens.

One major limitation of current post-decannulation care is that up to 25% of decannulated patients require reintubation within 7 days of decannulation.

The explanation for this is multifactorial and complex, with inadequate pulmonary rehabilitation being an important contributor.

During dressing-based management, patients are instructed to manually support the dressing during speech, coughing, or similar activities until the wound has healed-a period that may range from several days to weeks.

During the healing phase, airflow through the stoma may interfere with wound closure. In some patients, this leads to delayed healing and, in rare cases, to infection or the development of a chronic fistula between the trachea and the skin.

Previous attempts to seal the tracheostomy externally-from the skin side-have been associated with a high risk of subcutaneous emphysema, as air becomes trapped in the tissue between the trachea and the skin.

This type of treatment is therefore rarely used in clinical practice.

The New Treatment Concept In collaboration with a spin-out company from Aarhus University (IntraCair ApS), we have developed a concept that allows for intratracheal sealing of the tracheostomy.

In 2017, a previous research group at Aarhus University published the first study investigating such a sealing method in a porcine model.

Based on those experiments, we conducted a clinical feasibility study from 2020 to early 2022, in which a similar sealing disc was inserted in ICU patients, and immediate changes in lung physiology were measured.

These studies showed a marked improvement in both lung function and voice quality.

We have since advanced the concept and, in the period April-May 2022, tested our refined prototype in a porcine model.

By performing tracheostomy on nine pigs and inserting a disc constructed from medical-grade silicone, we demonstrated that the animals were able to ambulate and behave normally for 7 days while the disc provided intratracheal sealing.

The seal maintained airtightness under airway pressures equivalent to normal breathing and speech. However, some air leakage was observed under pressures corresponding to coughing.

In all nine pigs, the disc remained intact and correctly positioned throughout the observation period.

The disc is designed to be deconstructed by pulling on its "tail," allowing it to be removed without surgery through a nearly healed tracheostomy site. This removal method was successful in all cases.

In practice, it is not feasible to keep pigs under hygienically acceptable conditions for a full 7-day period.

To assess the biocompatibility of the chosen material, we therefore implanted the sealing disc in six pigs without placing it inside the trachea. Instead, the material was positioned externally on the trachea-isolated beneath the skin and without contact with the pigs' natural environment.

In all cases, normal physiological encapsulation of the material was observed, with no signs of adverse foreign body reaction.

Objective We aim to investigate our novel treatment method in patients with tracheostomies.

The study will evaluate the clinical applicability of the method and assess its effects on pulmonary function, phonation, and wound healing. Finally, we will explore whether the treatment has a beneficial impact on the rate of readmission among former ICU patients.

Study population A total of 35 participants from the Departments of Intensive Care and Otolaryngology - Head and Neck Surgery at Aarhus University Hospital will be included. All have previously undergone tracheostomy treatment.

Study Timeline Day -1 (the day before inclusion) Participants receive both oral and written information. A 24-hour reflection period is granted.

Day 0

Informed consent is signed by the participant. Decannulation is performed according to the department's standard procedure. Baseline assessments of voice and cough strength are conducted, along with spirometric measurement of pulmonary function.

The temporary intratracheal sealing disc is inserted into the tracheostomy tract. The disc is secured to the participant's neck using a dedicated fixation device.

Repeat measurements of voice, cough strength, and lung function are conducted. Photographic documentation of the tracheostomy site is obtained.

Day 1-6

Once daily, the following assessments are performed:

* Voice and cough strength
* Spirometry
* Photographic documentation of the tracheostomy site

Day 7 Final measurements of voice, cough strength, spirometry, and photographic documentation of the tracheostomy site are conducted.

The sealing disc is removed by gently pulling on the device's "tail" through the residual tracheostomy tract.

The participant is instructed to cough, and the site is observed for air leakage through the healed tracheostomy.

The participant completes a questionnaire designed in accordance with the SF-36 framework, to evaluate their experience with the sealing intervention.

If complete healing occurs prior to day 7, the sealing disc is removed earlier, and final assessments are conducted at that time.

Risks and Safety Measures

Four potential risks associated with the procedure have been identified:

Airway obstruction caused by the sealing disc. Irritation or infection of the tracheostomy site due to the sealing disc. Bleeding during insertion of the sealing disc. Accidental dislodgement of the sealing disc.

Ad 1: Airway obstruction Procedures conducted on day 1 will take place in the highly specialised ICU at Aarhus University Hospital under the supervision of a board-certified anaesthesiologist.

All standard airway management equipment will be immediately available. The procedure will be performed by Rasmus Ellerup Kraghede (MD, PhD fellow, Department of Cardiothoracic and Vascular Surgery) and Stig Dyrskog (Consultant, PhD, Department of Intensive Care).

Both have substantial experience with tracheostomy procedures and with the specific device used in this study.

Participants may experience a tickling sensation or mild discomfort in the airway during device insertion.

Insertion of the temporary sealing disc is expected to take less than 2 minutes.

To mitigate the risk of obstruction, the tail of the disc will be secured with a clamp during handling. Once in place, the tail will be fixed to the anterior neck so that the device cannot be dislodged without first being deconstructed and withdrawn through the tracheostomy tract.

For the entire 7-day intervention period, participants will be monitored continuously (24/7) by a dedicated member of the research team trained in airway management and emergency procedures related to the intervention.

If the participant is transferred to another ward, the observer will accompany the patient, and the study will continue in coordination with the receiving department.

In the unlikely event that the sealing device causes airway obstruction, appropriate emergency airway equipment will be available at the bedside at all times and will accompany the participant during any transfers.

The risk of airway obstruction has also been considered during the design phase. The average male tracheal cross-sectional area is approximately 2.8 cm². The sealing device has a thickness of 1.5 mm and a diameter of 26 mm, occupying at most one-third of the airway cross-section.

For comparison, tracheostomy tubes of size 7 and 8 occupy approximately 0.8 cm² and 1.1 cm², respectively, equivalent to one-third to one-half of the airway.

Due to the flexible nature of the silicone material, the disc conforms to the inner tracheal wall even in the presence of moderate displacing forces.

Ad 2: Irritation or infection The tracheostomy site will be inspected twice daily for signs of irritation or infection.

The sealing disc is made of medical-grade silicone, a well-established material used in implantable medical devices.

We consider the risk of a foreign body reaction to be very low, a conclusion supported by findings from our prior animal studies.

The sealing disc is manufactured by Technolution, an engineering company with expertise in the production of medical-grade silicone devices.

Sterile packaging is provided by the Central Sterile Supply Department at Aarhus University Hospital. Insertion and handling of the device will follow hospital protocols for sterility and hygiene in procedures related to tracheostomy.

Ad 3: Bleeding Theoretically, bleeding may occur during insertion of the sealing disc. This is considered a rare complication when manipulating a well-functioning tracheostomy.

Based on prior experience with the prototype, this complication was not observed in earlier clinical studies.

If unexpected bleeding occurs, in-room anaesthesia expertise will be available, and assistance from the Department of Otolaryngology can be summoned.

Overall, the risk is considered minimal.

Ad 4: Accidental dislodgement If the sealing disc is unintentionally dislodged, the participant will be in the same clinical situation as any other patient following decannulation.

We do not consider this event to represent any actual risk to the participant.

Data Protection All data will be handled in accordance with the Danish Data Protection Act and the General Data Protection Regulation (GDPR).

Participant data will be stored under anonymised participant ID numbers in the REDCap system, a recognised secure data management platform, ensuring controlled access and proper handling.

The principal investigator will maintain a separate list linking participant IDs to names and personal identification numbers. This list will be held exclusively by the principal investigator. All communications regarding participant data will use anonymised participant IDs only.

Signed consent forms will also be stored securely by the principal investigator.

Information Provided to Study Participants Potential participants will receive comprehensive oral and written information the day before removal of the tracheostomy tube (decannulation).

ELIGIBILITY:
Inclusion Criteria:

* Tracheostomy in place for ≥7 days for the purpose of mechanical ventilation in ICU
* Age ≥18 years
* Uncuffed or occluded tracheostomy tube (size 7-8) during the last 24 hours

Exclusion Criteria:

* Cognitive impairment or incapacity to such a degree that the participant is unable to comprehend study information or cooperate with the required assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-12-08 (Actual); Study Completion 2025-03-08 (Actual)

PRIMARY OUTCOMES:
Feasibilty | From inrollment to the end of treatment (maximum 7 days)
  Ease of device insertion, intratracheal placement, and removal will be assessed by the operating clinician immediately after each procedure. The evaluation will be based on a structured qualitative rating (easy, moderate, difficult) informed by the operator's direct experience and the patient's oral feedback during the procedure.The unit of measure will be the number of procedures rated in each category.
Patient satisfaction (Questionnaire-Based Score) | Filled out on the last day of dataretrieval (day 3-7)
  Patient satisfaction will be assessed using a structured questionnaire consisting of six items, each rated on a 5-point Likert scale (1 = very dissatisfied, 5 = very satisfied). Scores from individual items will be summarized by reporting the median (IQR) for each item across patients. The unit of measure will be the patient-reported score (range 1-5).

SECONDARY OUTCOMES:
Forced Vital Capacity (FVC) measured by spirometry | From enrollment and until removal of the device (up to 7 days after enrollment)
  Forced Vital Capacity (FVC) will be assessed by standard spirometry performed according to ATS/ERS guidelines. The unit of measure is liters (L). Measurement will be done daily. Results will be reported as median [IQR] or mean (SD) across patients.
Forced Expiratory Volume in 1 Second (FEV₁) measured by spirometry | From enrollment and until removal of the device (up to 7 days after enrollment)
  Forced Expiratory Volume in 1 Second (FEV₁) will be assessed by standard spirometry performed according to ATS/ERS guidelines. The unit of measure is liters (L). Measurement will be done daily. Results will be reported as median [IQR] or mean (SD).
Peak Expiratory Flow (PEF) measured by spirometry | From enrollment and until removal of the device (up to 7 days after enrollment)
  Peak Expiratory Flow (PEF) will be assessed by standard spirometry performed according to ATS/ERS guidelines. The unit of measure is liters/second (L/s). Measurement will be done daily. Results will be reported as median [IQR] or mean (SD).
Voice quality score | From enrollment and until removal of the device (up to 7 days after enrollment)
  Voice quality will be assessed from standardized patient voice recordings performed daily. Two trained professionals will independently rate overall clarity and strength of speech on a 6-point Likert scale (0 = inaudible, 5 = excellent). The unit of measure is the patient's mean voice quality score.
Tracheostomy wound healing status (photographic evaluation) | From enrollment and until removal of the device (up to 7 days after enrollment)
  Healing progression of the tracheostomy site will be assessed from standardized daily photographs evaluated by two independent clinicians. Wound status will be classified as incomplete, partial, or complete closure. The unit of measure will be the number and percentage of patients in each healing category at each assessment day.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark